CLINICAL TRIAL: NCT01381692
Title: A Randomized Phase I/II Study of Bortezomib, Rituximab, Dexamethasone and Temsirolimus in Patients With Relapsed Waldenstrom Macroglobulinemia and Relapsed/Refractory Mantle Cell, Follicular, Marginal Zone or Small Lymphocytic Lymphomas (Phase I), and Untreated/Relapsed Waldenstrom Macroglobulinemia (Phase II)
Brief Title: Bortezomib, Rituximab, and Dexamethasone With or Without Temsirolimus in Treating Patients With Untreated or Relapsed Waldenstrom Macroglobulinemia or Relapsed or Refractory Mantle Cell or Follicular Lymphoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2011-02650; NCI-2011-02650 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000701362; ECOG-E1A10; E1A10; E1A10 (Other: ECOG-ACRIN Cancer Research Group); E1A10 (Other: CTEP); U10CA180820 (NIH); U10CA021115 (NIH)
Record Dates: First submitted 2011-06-23; First posted 2011-06-27 (Estimated); Results first posted 2021-05-05 (Actual); Last update posted 2021-10-04 (Actual); Status verified 2021-09

CONDITIONS: Recurrent Follicular Lymphoma; Recurrent Mantle Cell Lymphoma; Recurrent Marginal Zone Lymphoma; Recurrent Non-Hodgkin Lymphoma; Recurrent Small Lymphocytic Lymphoma; Recurrent Waldenstrom Macroglobulinemia; Refractory Follicular Lymphoma; Refractory Mantle Cell Lymphoma; Refractory Marginal Zone Lymphoma; Refractory Non-Hodgkin Lymphoma; Refractory Small Lymphocytic Lymphoma
MeSH Terms: conditions — Lymphoma, Follicular; Lymphoma, Mantle-Cell; Lymphoma, B-Cell, Marginal Zone; Lymphoma, Non-Hodgkin; Leukemia, Lymphocytic, Chronic, B-Cell; Waldenstrom Macroglobulinemia | interventions — Bortezomib; Dexamethasone; Calcium Dobesilate; auricularum; dexamethasone acetate; dexamethasone 21-phosphate; Rituximab; CT-P10; temsirolimus; Sirolimus

ARMS (2):
- Arm I (rituximab, bortezomib, dexamethasone) (Active Comparator): Patients receive rituximab IV over 30-60 minutes on days 1, 8, 15, and 22 (of courses 1 and 4 only) and bortezomib IV or SC and dexamethasone PO on days 1, 8, and 15. Treatment repeats every 28 days for 6 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Bortezomib; Drug: Dexamethasone; Other: Laboratory Biomarker Analysis; Other: Quality-of-Life Assessment; Biological: Rituximab
- Arm II (temsirolimus, rituximab, bortezomib, dexamethasone) (Experimental): Patients receive temsirolimus IV over 30-60 minutes on days 1, 8, 15, and 22 and rituximab, bortezomib, and dexamethasone as in arm I. Treatment repeats every 28 days for 6 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Bortezomib; Drug: Dexamethasone; Other: Laboratory Biomarker Analysis; Other: Quality-of-Life Assessment; Biological: Rituximab; Drug: Temsirolimus

INTERVENTIONS:
Drug: Bortezomib — Given IV or SC
  Other Names: [(1R)-3-Methyl-1-[[(2S)-1-oxo-3-phenyl-2-[(pyrazinylcarbonyl)amino]propyl]amino]butyl]boronic Acid; LDP 341; MLN341; PS-341; PS341; Velcade
Drug: Dexamethasone — Given PO
  Other Names: Aacidexam; Adexone; Aknichthol Dexa; Alba-Dex; Alin; Alin Depot; Alin Oftalmico; Amplidermis; Anemul mono; Auricularum; Auxiloson; Baycadron; Baycuten; Baycuten N; Cortidexason; Cortisumman; Decacort; Decadrol; Decadron; Decadron DP; Decalix; Decameth; Decasone R.p.; Dectancyl; Dekacort; Deltafluorene; Deronil; Desamethasone; Desameton; Dexa-Mamallet; Dexa-Rhinosan; Dexa-Scheroson; Dexa-sine; Dexacortal; Dexacortin; Dexafarma; Dexafluorene; Dexalocal; Dexamecortin; Dexameth; Dexamethasone Intensol; Dexamethasonum; Dexamonozon; Dexapos; Dexinoral; Dexone; Dinormon; Dxevo; Fluorodelta; Fortecortin; Gammacorten; Hemady; Hexadecadrol; Hexadrol; Lokalison-F; Loverine; Methylfluorprednisolone; Millicorten; Mymethasone; Orgadrone; Spersadex; TaperDex; Visumetazone; ZoDex
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Biological: Rituximab — Given IV
  Other Names: ABP 798; BI 695500; C2B8 Monoclonal Antibody; Chimeric Anti-CD20 Antibody; CT-P10; IDEC-102; IDEC-C2B8; IDEC-C2B8 Monoclonal Antibody; MabThera; Monoclonal Antibody IDEC-C2B8; PF-05280586; Rituxan; Rituximab ABBS; Rituximab Biosimilar ABP 798; Rituximab Biosimilar BI 695500; Rituximab Biosimilar CT-P10; Rituximab Biosimilar GB241; Rituximab Biosimilar IBI301; Rituximab Biosimilar JHL1101; Rituximab Biosimilar PF-05280586; Rituximab Biosimilar RTXM83; Rituximab Biosimilar SAIT101; Rituximab Biosimilar SIBP-02; rituximab biosimilar TQB2303; rituximab-abbs; RTXM83; Truxima
Drug: Temsirolimus — Given IV
  Other Names: CCI-779; CCI-779 Rapamycin Analog; Cell Cycle Inhibitor 779; Rapamycin Analog; Rapamycin Analog CCI-779; Torisel
  Arms: Arm II (temsirolimus, rituximab, bortezomib, dexamethasone)

SUMMARY:
This randomized phase I/II trial studies the side effects and the best dose of temsirolimus when given together with bortezomib, rituximab, and dexamethasone and to see how well they work compared to bortezomib, rituximab, and dexamethasone alone in treating patients with untreated or relapsed Waldenstrom macroglobulinemia or relapsed or refractory mantle cell or follicular lymphoma. Bortezomib and temsirolimus may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Bortezomib may also stop the growth of cancer cells by blocking blood flow to the tumor. Monoclonal antibodies, such as rituximab, can block cancer growth in difference ways. Some block the ability of cancer cells to grow and spread. Others find cancer cells and help kill them or carry cancer-killing substances to them. Drugs used in chemotherapy, such as dexamethasone, work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. It is not yet known whether bortezomib, rituximab, and dexamethasone are more effective with temsirolimus in treating non-Hodgkin lymphoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the maximum tolerated dose (MTD) of temsirolimus in combination with bortezomib, rituximab, dexamethasone in patients with relapsed Waldenstrom's macroglobulinemia and relapsed/refractory mantle cell, follicular, marginal zone or small lymphocytic lymphoma. (Phase I) II. To evaluate whether the addition of temsirolimus to the regimen of bortezomib, rituximab, dexamethasone improves progression-free survival in patients with previously untreated or relapsed Waldenstrom's macroglobulinemia. (Phase II)

SECONDARY OBJECTIVES:

I. To define and describe the toxicities of temsirolimus in combination with bortezomib, rituximab, and dexamethasone. (Phase I) II. To evaluate time to progression of bortezomib, rituximab, dexamethasone +/- temsirolimus in patients. (Phase II) III. To evaluate major and minor response by 6 cycles of therapy of bortezomib, rituximab, dexamethasone +/- temsirolimus. (Phase II) IV. To evaluate time to response and duration of response of bortezomib, rituximab, dexamethasone +/- temsirolimus. (Phase II) V. To evaluate toxicity of bortezomib, rituximab, dexamethasone +/- temsirolimus. (Phase II) VI. To evaluate time to next therapy of bortezomib, rituximab, dexamethasone +/- temsirolimus. (Phase II) VII. To evaluate overall survival of bortezomib, rituximab, dexamethasone +/- temsirolimus. (Phase II) VIII. To describe treatment-related fatigue, physical and functional well-being during and after treatment. (Phase II) IX. To compare the change in treatment related fatigue, physical and functional well-being over 6 cycles of bortezomib, rituximab, dexamethasone +/- temsirolimus. (Quality of Life) X. To prospectively assess health-related quality of life longitudinally (pre-treatment to 3 year follow-up assessment) among trial participants. (Quality of Life) XI. To describe treatment-related peripheral neuropathy associated with bortezomib neurotoxicity. (Quality of Life)

OUTLINE: This is a phase I, dose-escalation study of temsirolimus followed by a randomized phase II study.

PHASE I: Patients receive temsirolimus intravenously (IV) over 30-60 minutes on days 1, 8, 15, and 22; rituximab IV over 30-60 minutes on days 1, 8, 15, and 22 (of courses 1 and 4 only); and bortezomib IV or subcutaneously (SC) and dexamethasone orally (PO) on days 1, 8, and 15. Courses repeat every 28 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.

PHASE II: Patients are randomized to 1 of 2 treatment arms.

ARM I: Patients receive rituximab IV over 30-60 minutes on days 1, 8, 15, and 22 (of courses 1 and 4 only) and bortezomib IV or SC and dexamethasone PO on days 1, 8, and 15. Treatment repeats every 28 days for 6 courses in the absence of disease progression or unacceptable toxicity.

ARM II: Patients receive temsirolimus IV over 30-60 minutes on days 1, 8, 15, and 22 and rituximab, bortezomib, and dexamethasone as in arm I. Treatment repeats every 28 days for 6 courses in the absence of disease progression or unacceptable toxicity.

After completion of study therapy, patients are followed up every 3 months for 2 years, every 6 months for 3 years, and then yearly for 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven diagnosis
* For phase I portion (Arm A, B, C and D), patients must have of one of the following:

  * Relapsed Waldenstrom's macroglobulinemia
  * Relapsed/refractory mantle cell lymphoma; previous treatment with at least one standard regimen and no longer responsive to that regimen
  * Relapsed/refractory follicular lymphoma; previous treatment with at least one standard regimen and no longer responsive to that regimen
  * Relapsed/refractory marginal zone lymphoma; previous treatment with at least one standard regimen and no longer responsive to that regimen
  * Relapsed/refractory small lymphocytic lymphoma; previous treatment with at least one standard regimen and no longer responsive to that regimen
* For phase II portion (Arm E and F), patients must have a diagnosis of symptomatic Waldenstrom's macroglobulinemia, either untreated or relapsed, confirmed by the presence of all of the following:

  * Bone marrow lymphoplasmacytosis with

    * >= 10% lymphoplasmatic cells (measured within 28 days prior to registration) OR
    * Aggregates or sheets of one of the following: lymphocytes, plasma cells or lymphoplasmacytic cells on the bone marrow biopsy (measured within 28 days prior to registration)
  * Measurable disease defined as a quantitative immunoglobulin M (IgM) monoclonal protein of >= 1000 mg/dL obtained within 28 days prior to registration
  * Cluster of differentiation 20 (CD20) positive bone marrow or lymph node by immunohistochemistry or flow cytometry obtained within 28 days prior to registration
  * Lymph node biopsy must be done =< 28 days prior to registration if used as an eligibility criterion for study entry
  * Serum protein electrophoresis (SPEP) is required to be performed within 28 days prior to registration
* Additional requirements for Waldenstrom's macroglobulinemia (WM) patients (phase I and II):
* In addition to measurable disease, patients must have symptomatic disease defined by one or more of the following:

  * Laboratory studies defining eligibility (hemoglobin [Hgb], platelet count, viscosity) must have been obtained within 28 days prior to registration; if more than one test was obtained, the most recent one will be utilized
  * Hemoglobin =< 11 g/dL
  * Hyperviscosity syndrome or measured viscosity level of >= 4 centipoise

    * NOTE: for these patients it is strongly recommended that they undergo therapeutic plasmapheresis prior to initiation of therapy
  * Platelet count < 100,000/mm^3
  * Symptomatic lymphadenopathy, splenomegaly, or hepatomegaly
  * Constitutional symptoms including fever, night sweats, or unexplained weight loss (at least 10% of body weight in < 6 months)
  * Symptomatic cryoglobulinemia
* Additional requirements for WM patients (phase I):

  * Patients must have received previous treatment with at least one standard regimen and are no longer responsive to that regimen
  * There must have been at least 21 days since the last regimen and patient must have recovered from any previous treatment-related toxicity to =< grade 1
* Additional requirements for WM patients (phase II):

  * For previously treated patients, no more than 4 prior regimens are allowed
  * If last regimen is with rituximab there must have been at least 6 months since last rituximab dose, and if without rituximab there must have been at least 3 months since last regimen
* For all phase I patients, there must have been at least 21 days since last regimen and any previous non-hematologic treatment related toxicity must have resolved to =< grade 1
* Patients must not be receiving concurrent steroids > 10 mg prednisone (or equivalent) per day
* Prior irradiation is allowed if >= 28 days prior to registration have elapsed since the date of last treatment
* Fasting serum cholesterol =< 300 mg/dL OR =< 7.75 mmol/L AND fasting triglycerides =< 2.5 x institutional upper limit of normal (ULN), within 28 days prior to registration

  * NOTE: in case one or both of these thresholds are exceeded, the patient can only be included after initiation of appropriate lipid lowering medication; patients cannot be enrolled if they do not meet these criteria on or off lipid lowering medication; patients must start lipid lowering medication and cholesterol and triglycerides must be below said levels before study entry
* Patients must not have had prior exposure to mammalian target of rapamycin (m-TOR) inhibitors (sirolimus, temsirolimus, everolimus)
* Women must not be pregnant or breast-feeding; all females of childbearing potential must have a blood test or urine study within 2 weeks prior to registration to rule out pregnancy; a female of childbearing potential is any woman, regardless of sexual orientation or whether they have undergone tubal ligation, who meets the following criteria: 1) has not undergone a hysterectomy or bilateral oophorectomy; or 2) has not been naturally postmenopausal for at least 24 consecutive months (i.e., has had menses at any time in the preceding 24 consecutive months)
* Women of childbearing potential and sexually active males must use an accepted and effective method of contraception throughout the study and for 8 weeks following discontinuation of everolimus
* Patients must have no history of prior malignancy except for adequately treated basal cell or squamous cell skin cancer or in-situ cervical cancer; the patient may also have had other cancer for which the patient was curatively treated with surgery alone and from which the patient has been disease free for >= 5 years
* Platelets >= 75,000 mm^3
* Neutrophils >= 1,000 mm^3
* Serum glutamic oxaloacetic transaminase (SGOT) (aspartate aminotransferase [AST]) and serum glutamate pyruvate transaminase (SGPT) (alanine aminotransferase [ALT]) =< 2.5 x institutional ULN
* Direct bilirubin =< 1.5 mg/dL
* Serum creatinine =< 2.5 mg/dL
* Patients must be tested for hepatitis B surface antigen (HBsAg) and hepatitis B core antibody (anti-HBc) within 28 days of registration and will not be eligible if found to be positive
* Patients must not have any severe and/or uncontrolled medical condition or other conditions that could affect their participation in the study, including, but not restricted to:

  * Symptomatic congestive heart failure of New York Heart Association class III or IV
  * Unstable angina pectoris, symptomatic congestive heart failure, myocardial infarction within 3 months of start of study treatment, serious uncontrolled cardiac arrhythmia or any other clinically significant heart disease
  * Severely impaired lung function as defined as spirometry and diffusing capacity of the lung for carbon monoxide (DLCO) (corrected for Hgb) that is < 50% of the normal predicted value and/or oxygen (O2) saturation < 88% at rest on room air
  * Active (acute or chronic) or uncontrolled severe infections
* Patients must have Eastern Cooperative Oncology Group (ECOG)-American College of Radiology Imaging Network (ACRIN) performance status of =< 2
* Patients must not have grade 2 or higher neuropathy
* Patients must not have concurrent use of angiotensin-converting enzyme (ACE) inhibitors (angioedema), and no concurrent use of strong cytochrome P450, family 3, subfamily A, polypeptide 4 (CYP3A4) inducers and inhibitors

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2011-07-20 (Actual); Primary Completion 2014-12-08 (Actual); Study Completion 2021-09-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Leonard T Heffner, Principal Investigator — ECOG-ACRIN Cancer Research Group
Locations (11):
- United States (11):
  - Presbyterian - Saint Lukes Medical Center - Health One, Denver, Colorado
  - Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Geisinger Medical Center, Danville, Pennsylvania
  - University of Pennsylvania/Abramson Cancer Center, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - Marshfield Medical Center-Marshfield, Marshfield, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
  - Marshfield Clinic-Minocqua Center, Minocqua, Wisconsin

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All patients were accrued between July 20, 2011 and August 15, 2014.
Groups:
- Arm A (Phase I: Temsirolimus Dose Level 1, Rituximab, Bortezomib, Dexamethasone): Patients receive temsirolimus IV at dose level 1 over 30-60 minutes on days 1, 8, 15, and 22, rituximab IV over 30-60 minutes on days 1, 8, 15, and 22 (of courses 1 and 4 only), bortezomib IV or SC and dexamethasone PO on days 1, 8, and 15. Treatment repeats every 28 days for 6 courses in the absence of disease progression or unacceptable toxicity.
- Arm B (Phase I: Temsirolimus Dose Level 2, Rituximab, Bortezomib, Dexamethasone): Patients receive temsirolimus IV at dose level 2 over 30-60 minutes on days 1, 8, 15, and 22, rituximab IV over 30-60 minutes on days 1, 8, 15, and 22 (of courses 1 and 4 only), bortezomib IV or SC and dexamethasone PO on days 1, 8, and 15. Treatment repeats every 28 days for 6 courses in the absence of disease progression or unacceptable toxicity.
- Arm C (Phase I: Temsirolimus Dose Level 3, Rituximab, Bortezomib, Dexamethasone): Patients receive temsirolimus IV at dose level 3 over 30-60 minutes on days 1, 8, 15, and 22, rituximab IV over 30-60 minutes on days 1, 8, 15, and 22 (of courses 1 and 4 only), bortezomib IV or SC and dexamethasone PO on days 1, 8, and 15. Treatment repeats every 28 days for 6 courses in the absence of disease progression or unacceptable toxicity.
- Arm D (Phase I: Temsirolimus Dose Level 4, Rituximab, Bortezomib, Dexamethasone): Patients receive temsirolimus IV at dose level 4 over 30-60 minutes on days 1, 8, 15, and 22, rituximab IV over 30-60 minutes on days 1, 8, 15, and 22 (of courses 1 and 4 only), bortezomib IV or SC and dexamethasone PO on days 1, 8, and 15. Treatment repeats every 28 days for 6 courses in the absence of disease progression or unacceptable toxicity.
- Arm E (Phase II: Rituximab, Bortezomib, Dexamethasone): Patients receive rituximab IV over 30-60 minutes on days 1, 8, 15, and 22 (of courses 1 and 4 only) and bortezomib IV or SC and dexamethasone PO on days 1, 8, and 15. Treatment repeats every 28 days for 6 courses in the absence of disease progression or unacceptable toxicity.
- Arm F (Phase II: Temsirolimus, Rituximab, Bortezomib, Dexamethasone): Patients receive temsirolimus IV over 30-60 minutes on days 1, 8, 15, and 22 and rituximab, bortezomib, and dexamethasone as in arm E. Treatment repeats every 28 days for 6 courses in the absence of disease progression or unacceptable toxicity.
Period: Overall Study
Arm/Group | Arm A (Phase I: Temsirolimus Dose Level 1, Rituximab, Bortezomib, Dexamethasone) | Arm B (Phase I: Temsirolimus Dose Level 2, Rituximab, Bortezomib, Dexamethasone) | Arm C (Phase I: Temsirolimus Dose Level 3, Rituximab, Bortezomib, Dexamethasone) | Arm D (Phase I: Temsirolimus Dose Level 4, Rituximab, Bortezomib, Dexamethasone) | Arm E (Phase II: Rituximab, Bortezomib, Dexamethasone) | Arm F (Phase II: Temsirolimus, Rituximab, Bortezomib, Dexamethasone)
Started | 7 | 2 | 0 | 0 | 0 | 0
Completed | 6 | 2 | 0 | 0 | 0 | 0
Not Completed | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 1 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All patients enrolled are included in this analysis.
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A (Phase I: Temsirolimus Dose Level 1, Rituximab, Bortezomib, Dexamethasone) | Arm B (Phase I: Temsirolimus Dose Level 2, Rituximab, Bortezomib, Dexamethasone) | Total
Number analyzed (Participants) | 7 | 2 | 9
Age, Continuous [Median (Full Range); unit: years] | 61 [47 to 82] | 72 [64 to 80] | 64 [47 to 82]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 3
  Male | 5 | 1 | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 7 | 2 | 9
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 6 | 2 | 8
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Phase I: The Maximum Tolerated Dose (MTD) of Temsirolimus in Combination With Bortezomib, Rituximab and Dexamethasone
Description: Temsirolimus in combination with bortezomib, rituximab, dexamethasone were to be escalated using a standard 3+3 design. The MTD was defined as the highest dose level at which no more than 0 in 3 or 1 in 6 participants experienced a dose-limiting toxicity (DLT) during the first 28-day cycle of treatment.
Time Frame: Assessed during cycle 1 (28 days)
Measure: Number; unit: mg
Arm/Group | Arm A (Phase I: Temsirolimus Dose Level 1, Rituximab, Bortezomib, Dexamethasone) | Arm B (Phase I: Temsirolimus Dose Level 2, Rituximab, Bortezomib, Dexamethasone)
Number analyzed (Participants) | 7 | 2
mg | NA — The maximum tolerated dose (MTD) of temsirolimus was not determined because the study was terminated early due to slow accrual. | NA — The maximum tolerated dose (MTD) of temsirolimus was not determined because the study was terminated early due to slow accrual.

2. Primary Outcome: Phase II: Progression-free Survival
Description: Progression-free survival is defined as the time from randomization to progression or death, whichever occurred first.
  Progression is evaluated based on Recommended Response Criteria for Waldenstrom's Macroglobulinemia. Progression is defined as at least 25% increase in serum monoclonal IgM protein by electrophoresis confirmed by a second measurement at any time, as well as an absolute increase of the M-spike by 0.5g/dL, or progression of clinically significant findings due to disease, (i.e. anemia, thrombocytopenia, leukopenia, bulky adenopathy/organomegaly or symptoms of disease) or hyperviscosity, neuropathy, symptomatic cryoglobulinemia, or amyloidosis attributable to WM.
Time Frame: Assessed every 3 months if <2 years from study entry, every 6 months if 2-5 years from study entry, and annually if 6-10 years
Population: No patients were enrolled in the phase II part of this study.
Arm/Group | Arm E (Phase II: Rituximab, Bortezomib, Dexamethasone) | Arm F (Phase II: Temsirolimus, Rituximab, Bortezomib, Dexamethasone)
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Phase II: Time to Progression
Description: Time to progression is defined as the time from randomization to disease progression.
  Progression is evaluated based on Recommended Response Criteria for Waldenstrom's Macroglobulinemia. Progression is defined as at least 25% increase in serum monoclonal IgM protein by electrophoresis confirmed by a second measurement at any time, as well as an absolute increase of the M-spike by 0.5g/dL, or progression of clinically significant findings due to disease, (i.e. anemia, thrombocytopenia, leukopenia, bulky adenopathy/organomegaly or symptoms of disease) or hyperviscosity, neuropathy, symptomatic cryoglobulinemia, or amyloidosis attributable to WM.
Time Frame: as for outcome 2
Population: No patients were enrolled in the phase II part of this study.
Arm/Group | Arm E (Phase II: Rituximab, Bortezomib, Dexamethasone) | Arm F (Phase II: Temsirolimus, Rituximab, Bortezomib, Dexamethasone)
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Phase II: Major Response Rate
Description: Response is evaluated based on Recommended Response Criteria for Waldenstrom's Macroglobulinemia (WM). Major response is defined as complete response (CR), near CR (nCR), very good partial remission (VGPR), or partial response (PR).
  CR: Disappearance of monoclonal protein by immmunofixation; no histologic evidence of bone marrow involvement, resolution of any adenopathy/organomegaly, or signs or symptoms attributable to WM Near CR (nCR): As for CR except that immunofixation is still positive VGPR: At least 90% reduction of serum monoclonal protein using serum protein electrophoresis (SPEP) PR: At least 50% reduction of serum monoclonal concentration on protein electrophoresis and at least a decrease in adenopathy/organomegaly (confirmed by original mode of imaging). No new signs or symptoms of active disease.
Time Frame: Assessed at cycle 6
Population: No patients were enrolled in the phase II part of this study.
Arm/Group | Arm E (Phase II: Rituximab, Bortezomib, Dexamethasone) | Arm F (Phase II: Temsirolimus, Rituximab, Bortezomib, Dexamethasone)
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Phase II: Minor Response Rate
Description: Response is evaluated based on Recommended Response Criteria for Waldenstrom's Macroglobulinemia (WM). Minor response is defined as achieving minor response (MR) or better (including complete response [CR], near CR (nCR), very good partial remission [VGPR], partial response [PR] and MR).
  CR: Disappearance of monoclonal protein by immmunofixation; no histologic evidence of bone marrow involvement, resolution of any adenopathy/organomegaly, or signs or symptoms attributable to WM nCR: As CR except that immunofixation is still positive VGPR: At least 90% reduction of serum monoclonal protein using serum protein electrophoresis PR: At least 50% reduction of serum monoclonal concentration on protein electrophoresis and at least a decrease in adenopathy/organomegaly (confirmed by original mode of imaging). No new signs or symptoms of active disease.
  MR: At least 25% but less than 50% reduction of serum monoclonal protein and no new signs or symptoms of active disease.
Time Frame: Assessed at cycle 6
Population: No patients were enrolled in the phase II part of this study.
Arm/Group | Arm E (Phase II: Rituximab, Bortezomib, Dexamethasone) | Arm F (Phase II: Temsirolimus, Rituximab, Bortezomib, Dexamethasone)
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Phase II: Time to Response
Description: Time to response is defined as the time from randomization to documentation of response. Response is evaluated based on Recommended Response Criteria for Waldenstrom's Macroglobulinemia (WM). Response is defined as complete response (CR), near CR (nCR), very good partial remission (VGPR), partial response (PR) or minor response (MR).
  CR: Disappearance of monoclonal protein by immmunofixation; no histologic evidence of bone marrow involvement, resolution of any adenopathy/organomegaly, or signs or symptoms attributable to WM nCR: As CR except that immunofixation is still positive VGPR: >=90% reduction of serum monoclonal protein using serum protein electrophoresis PR: >=50% reduction of serum monoclonal concentration on protein electrophoresis and at least a decrease in adenopathy/organomegaly (confirmed by original mode of imaging). No new signs or symptoms of active disease.
  MR: >=25% but <50% reduction of serum monoclonal protein. No new signs or symptoms of active disease
Time Frame: Assessed every 3 months if <2 years of study entry, every 6 months if 2-5 years of study entry, and annually if 6-10 years
Population: No patients were enrolled in the phase II part of this study.
Arm/Group | Arm E (Phase II: Rituximab, Bortezomib, Dexamethasone) | Arm F (Phase II: Temsirolimus, Rituximab, Bortezomib, Dexamethasone)
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Phase II: Duration of Response
Description: Duration of response is defined as the time from documentation of response to disease progression. Response evaluation will be based on the Recommended Response Criteria for Waldenstrom's Macroglobulinemia (WM).
  Response is defined as complete response (CR), near CR (nCR), very good partial remission (VGPR), partial response (PR) or minor response (MR). Progression is defined as at least 25% increase in serum monoclonal IgM protein by electrophoresis confirmed by a second measurement at any time, as well as an absolute increase of the M-spike by 0.5g/dL, or progression of clinically significant findings due to disease, or hyperviscosity, neuropathy, symptomatic cryoglobulinemia, or amyloidosis attributable to WM.
Time Frame: as for outcome 6
Population: No patients were enrolled in the phase II part of this study.
Arm/Group | Arm E (Phase II: Rituximab, Bortezomib, Dexamethasone) | Arm F (Phase II: Temsirolimus, Rituximab, Bortezomib, Dexamethasone)
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Phase II: Time to Next Therapy
Description: Time to next therapy is defined as duration from the end of protocol treatment to the initiation of next therapy, censored at date last known alive without initiation of next therapy.
Time Frame: as for outcome 6
Population: No patients were enrolled in the phase II part of this study.
Arm/Group | Arm E (Phase II: Rituximab, Bortezomib, Dexamethasone) | Arm F (Phase II: Temsirolimus, Rituximab, Bortezomib, Dexamethasone)
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Phase II: Overall Survival
Description: Overall survival is defined as the time from randomization to date of death or date last known alive.
Time Frame: as for outcome 6
Population: No patients were enrolled in the phase II part of this study.
Arm/Group | Arm E (Phase II: Rituximab, Bortezomib, Dexamethasone) | Arm F (Phase II: Temsirolimus, Rituximab, Bortezomib, Dexamethasone)
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Assessed every 4 weeks while on treatment and for 30 days after the end of treatment
Arm/Group | Arm A (Phase I: Temsirolimus Dose Level 1, Rituximab, Bortezomib, Dexamethasone) | Arm B (Phase I: Temsirolimus Dose Level 2, Rituximab, Bortezomib, Dexamethasone)
All-Cause Mortality (participants affected / at risk) | 1/7 | 0/2
Serious Adverse Events (participants affected / at risk) | 7/7 | 1/2
Other Adverse Events (participants affected / at risk) | 7/7 | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A (Phase I: Temsirolimus Dose Level 1, Rituximab, Bortezomib, Dexamethasone) (N=7) | Arm B (Phase I: Temsirolimus Dose Level 2, Rituximab, Bortezomib, Dexamethasone) (N=2)
Anemia (Blood and lymphatic system disorders) | 1 | 0
Diarrhea (Gastrointestinal disorders) | 3 | 0
Nausea (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0
Lymphocyte count decreased (Investigations) | 1 | 0
Neutrophil count decreased (Investigations) | 3 | 1
Platelet count decreased (Investigations) | 3 | 0
White blood cell decreased (Investigations) | 2 | 1
Hyperglycemia (Metabolism and nutrition disorders) | 1 | 0
Hypertriglyceridemia (Metabolism and nutrition disorders) | 2 | 0
Hypokalemia (Metabolism and nutrition disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A (Phase I: Temsirolimus Dose Level 1, Rituximab, Bortezomib, Dexamethasone) (N=7) | Arm B (Phase I: Temsirolimus Dose Level 2, Rituximab, Bortezomib, Dexamethasone) (N=2)
Anemia (Blood and lymphatic system disorders) | 5 | 1
Edema limbs (General disorders) | 3 | 0
Fatigue (General disorders) | 5 | 1
Localized edema (General disorders) | 1 | 0
Pain (General disorders) | 2 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 0
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 | 0
Constipation (Gastrointestinal disorders) | 2 | 0
Diarrhea (Gastrointestinal disorders) | 5 | 0
Mucositis oral (Gastrointestinal disorders) | 3 | 1
Nausea (Gastrointestinal disorders) | 1 | 1
Lung infection (Infections and infestations) | 1 | 0
Nail infection (Infections and infestations) | 1 | 0
Sinusitis (Infections and infestations) | 1 | 1
Skin infection (Infections and infestations) | 0 | 1
Upper respiratory infection (Infections and infestations) | 1 | 0
Bruising (Injury, poisoning and procedural complications) | 1 | 0
Alanine aminotransferase increased (Investigations) | 3 | 0
Alkaline phosphatase increased (Investigations) | 1 | 1
Aspartate aminotransferase increased (Investigations) | 3 | 0
Blood bilirubin increased (Investigations) | 1 | 0
Cholesterol high (Investigations) | 4 | 1
Creatinine increased (Investigations) | 1 | 0
Lymphocyte count decreased (Investigations) | 3 | 1
Neutrophil count decreased (Investigations) | 7 | 1
Platelet count decreased (Investigations) | 6 | 1
White blood cell decreased (Investigations) | 7 | 1
Investigations - Other, specify (Investigations) | 1 | 0
Anorexia (Metabolism and nutrition disorders) | 2 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 4 | 2
Hypertriglyceridemia (Metabolism and nutrition disorders) | 5 | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 | 0
Hypocalcemia (Metabolism and nutrition disorders) | 1 | 0
Hypokalemia (Metabolism and nutrition disorders) | 1 | 0
Hyponatremia (Metabolism and nutrition disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
Dizziness (Nervous system disorders) | 1 | 0
Dysgeusia (Nervous system disorders) | 1 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 1 | 0
Insomnia (Psychiatric disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Urinary frequency (Renal and urinary disorders) | 0 | 1
Flushing (Vascular disorders) | 1 | 0
Hot flashes (Vascular disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less